CLINICAL TRIAL: NCT00452725
Title: Effect of the Growth Hormone MAXOMAT ® on the Growth of Small Children and Adolescents (<-2 SD) Due to NOONAN's Syndrome
Brief Title: Effect of MAXOMAT ® on the Growth of Small Children to NOONAN's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAX08
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Noonan Syndrome
MeSH Terms: conditions — Noonan Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MAXOMAT ®, biosynthetic growth hormone — 2 posologies according to age (children and adolescents) treatment is planned for a 2 year duration

SUMMARY:
1. Clinical Objective : To improve the growth of these children
2. Genetic objective : A study of the genetics of the syndrome

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with Noonan's syndrome with a height < -2 SD and no progressive cardiopathy

Exclusion Criteria:

* Age < 3 years
* Height ≥ -2 SD

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 1997-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of height : gain in height and rate of growth | at each visit (every 3 months) or every 6 months

SECONDARY OUTCOMES:
Clinical and laboratory test safety | every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France